CLINICAL TRIAL: NCT06729450
Title: Split-face Efficacy and Tolerability of DispersinB Acne Cleanser in the Treatment of Mild to Moderate Acne Vulgaris
Brief Title: Efficacy and Tolerability of DispersinB Acne Cleanser in the Treatment of Mild to Moderate Acne Vulgaris
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kane Biotech Inc (Industry)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB-A001
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Acne Vulgaris on the Face
Keywords: acne; dermatosis
MeSH Terms: conditions — Acne Vulgaris; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- intra-individual Split-face comparison (Experimental): Subjects will complete baseline assessments and be randomized (left face versus right face) to apply DispersinB Acne Cleanser over at 12-week treatment period, for an intra-individual, split-face comparison. Subjects will use the DispersinB Acne Cleanser on the assigned facial side for 5 minutes and then will use the provided 4% Benzoyl peroxide facial wash to wash entire face for daily (evening) use.
  Interventions: Device: DispersinB Acne Cleanser

INTERVENTIONS:
Device: DispersinB Acne Cleanser — DispersinB Acne Cleanser, strength: 80 ug/g, topical gel

SUMMARY:
This is a single-center study using intra-individual comparison (right half-face versus left half-face) to evaluate the efficacy and tolerability of DispersinB Acne Cleanser for treatment of acne in adults. An initial sample size of 24 subjects is planned to be randomized in order to provide proof of concept efficacy and tolerability of the product.

The main questions it aims to answer are:

1. Percent of subjects rated "Clear" and "Almost Clear" on a 5-point scale 0=clear; 4=severe) at 12 weeks
2. Change in inflammatory and noninflammatory lesion count per half-face at 12 weeks

Researchers will compare each half-face:

* one half facial wash with DispersinB Acne Cleanser and 4% Benzoyl Peroxide.
* one half facial wash with 4% Benzoyl Peroxide only

Subjects will use the DispersinB Acne Cleanser on the assigned facial side for 5 minutes and then will use the provided 4% Benzoyl peroxide facial wash to wash entire face for daily (evening) use.

DETAILED DESCRIPTION:
This is a single-center study using intra-individual comparison (right half-face versus left half-face) to evaluate the efficacy and tolerability of DispersinB Acne Cleanser for treatment of acne. An initial sample size of 24 subjects is planned to be randomized in order to provide proof of concept efficacy and tolerability of the product.

Subject eligibility is evaluated over a 28-day screening period. Qualified subjects will complete baseline assessments and be randomized (left face versus right face) to apply DispersinB Acne Cleanser over at 12-week treatment period, for an intra-individual, split-face comparison. Subjects will use the DispersinB Acne Cleanser on the assigned facial side for 5 minutes and then will use the provided 4% Benzoyl peroxide facial wash to wash entire face for daily (evening) use.

Subjects who do not require a washout period may complete the Screening and Baseline visit/assessments on the same day. Subjects who initially fail screening may be re-screened once.

Subjects will return to the clinic for efficacy and tolerability assessments at weeks 2, 4, 8, and 12. Study procedures and assessments are performed according to the schedule of activities, Section 1.3.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 18 years or older, at screening visit.
2. Subject with clinical diagnosis of acne vulgaris on the face as defined by Investigator's Global Assessment (IGA) score of 2 (Mild) or 3 (Moderate), with the same score on both sides of the face.
3. Subject with a symmetrical number of lesions on the whole face.
4. The subject is a female of childbearing potential is willing to undergo UPTs throughout the study.
5. Subject having read, understood, and signed the approved Informed Consent Form (ICF) prior to any participation in the study.
6. Subject agrees and is able to comply with all time commitments and procedural requirements of the protocol.
7. Subject agrees to having facial photographs taken and verified by the subject signing an approved photography ICF.
8. Subject is informed of terms pertaining to personal information protection and privacy and is willing to share personal information and data, as verified by signing a written authorization form.

Exclusion Criteria:

1. Subject with acne types other than acne vulgaris.
2. Subject with dermal conditions on the face that may interfere with study assessments in the opinion of the investigator (tattoo, skin abrasion, eczema, sun burn, scars, large nevi, etc.).
3. Subject with excessive facial hair that would interfere with study assessments, as judged by the investigator.
4. Pregnant women (positive urine pregnancy test at screening or baseline) or women planning pregnancy during the study.
5. Subjects taking Vitamin A supplements in excess of the recommended daily allowance (4000-5000 IU; no washout period is required).
6. Subject with a washout period for topical treatment or procedures on the face less than:

   1. Topical treatments: corticosteroids, antibiotics, azelaic acid, alpha hydroxy acids, salicylic acid, zinc containing treatments, hydroquinones, and other anti-acne treatments - 2 weeks
   2. Topical retinoids - 2 weeks
   3. Calascoterone cream 1% - 2 weeks
   4. Cosmetic/aesthetic procedures (e.g., comedo extraction, desquamating, or abrasive agents, adhesive "pore" cleansing strips) - 1 week
   5. Wax epilation - 2 weeks
   6. Photodynamic therapy - 4 weeks
   7. Laser therapy, microdermabrasion, deep chemical peel, and other plastic surgical treatments for acne - 12weeks
7. Subject with a washout period for systemic treatment less than:

   1. Corticosteroids (except locally acting such as inhaled or intrathecal), antibiotics, and spironolactone - 4 weeks
   2. Oral retinoids/isotretinoin - 12 weeks
   3. Cyproterone acetate/Chlomadinone acetate - 12 weeks
   4. Immunomodulators - 12 weeks
8. Subject is currently receiving any prescription testosterone therapy or on a testosterone booster or supplements.
9. The subject is unwilling or unable to refrain from use of prohibited medication or procedures during the study.
10. Subject who will experience intensive ultraviolet exposure during the study (sunbathing, tanning beds, etc.).
11. Subject with an acute/chronic disease or a history of major medical, surgical, or psychiatric condition or surgical interventions that may interfere with the interpretation of the study results.
12. Study site personnel or employees/close relatives of the study Sponsor.
13. Subject who has participated in another investigational treatment study within 30 days prior to screening.
14. Subject with a history of alcohol/drug abuse.
15. Subject who is unable to communicate or cooperate with the investigator due to language problems or impaired cognitive/verbal function.
16. Subject is currently incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Success rate per half-face | Baseline to week 12
  Success rate per half-face on the Investigator's Global Assessment - Percent of subjects rated "Clear" and "Almost Clear" on a 5-point scale (0=clear; 4=severe)
Change in inflammatory and noninflammatory lesion count | baseline to week 12
  Change in inflammatory and noninflammatory lesion count per half-face - change in lesion counts equals week 12 count minus baseline count

SECONDARY OUTCOMES:
Local tolerability | baseline to week 12
  Local tolerability parameters (erythema, scaling, dryness, and stinging/burning) will be evaluated per half-face - Worst post-baseline assessment rated on a 5-point scale (0=none; 4=strong)

CONTACTS AND LOCATIONS:
Overall Officials: Prinicipal Investigator, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No